CLINICAL TRIAL: NCT04136769
Title: Preoperative/Neoadjuvant Therapy and Vascular Debranching Followed by Resection for Locally Advanced Pancreatic Cancer
Acronym: PREVADER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Substantial delays in recruitment
Sponsor: Ulrich Ronellenfitsch, MD (Other)
Responsible Party: Sponsor-Investigator, Ulrich Ronellenfitsch, MD, Study Coordinator, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-152
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Pancreas Cancer
Keywords: Arterial Invasion; Arterial reconstruction; Neoadjuvant chemotherapy; Tumor resection
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Exact single stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): After trial enrolment, patients undergo visceral debranching.
  After visceral debranching, patients proceed to neoadjuvant chemotherapy. The therapy as such is not a formal part of the trial protocol. The specific chemotherapy regimen and its duration are decided individually by treating physicians.
  Tumor resection should be performed two to four weeks after completion of chemotherapy. Prior to resection, re-staging and verification of vascular reconstruction patency are carried out. The specific procedure for tumor resection and intestinal tract reconstruction is at the choice of the treating surgeon. It should follow oncological principles and aim at complete removal of the tumor and regional lymph nodes. Usually, resection will be done as pancreatoduodenectomy with or without distal gastrectomy (Whipple's procedure or pylorus-preserving Whipple's procedure), distal pancreatectomy with splenectomy, or total pancreatectomy with splenectomy.
  Interventions: Procedure: Visceral Debranching

INTERVENTIONS:
Procedure: Visceral Debranching — Visceral debranching is defined as a vascular reconstruction with the aim of ensuring a sufficient arterial blood flow to the mesentery and liver after the subsequently planned tumor resection, which usually comprises ligation of the gastroduodenal artery or other relevant collateral vessels. All open vascular procedures can be employed for visceral debranching. Examples are aorto-visceral or iliaco-visceral bypasses using autologous vein or an allogeneic graft, or re-insertion of the superior mesenteric artery or celiac trunk into the aorta.
  Other Names: Revascularisation of visceral arteries

SUMMARY:
Pancreatic cancer continues to have a poor prognosis. Many patients are diagnosed with advanced disease. In a considerable proportion of these patients, the tumor has contact with or invades into arterial blood vessels supplying the liver or bowel. Moreover, some patients have anatomical variations or Stenosis of these vessels. All such cases require a surgical reconstruction of the blood vessels upon pancreatic cancer resection in order to prevent that the liver or bowel are not sufficiently supplied with blood anymore. Performing such arterial reconstruction in one operation along with tumor resection is associated with a relevant risk of complications or even death.

This trial evaluates if the approach of 'visceral debranching', i.e. surgical reconstruction of arterial blood vessels supplying the liver or bowel, prior to chemotherapy and finally tumor resection in patients with locally advanced pancreatic cancer, is feasible.

ELIGIBILITY:
Inclusion Criteria

* Pancreatic cancer (pancreatic ductal adenocarcinoma, Intraductal papillary mucinous neoplasm (IPMN) - derived adenocarcinoma, adenosquamous carcinoma), diagnosed by preoperative biopsy or cytology or intraoperative biopsy during the visceral debranching procedure
* Evidence of locally advanced disease which is considered unresectable due to arterial invasion on CT or MRI according to National Comprehensive Cancer Network (NCCN) and International Study Group of Pancreatic Surgery (ISGPS) criteria:

  * Tumor encasement (>180°) of the superior mesenteric artery or celiac trunk
  * Tumor encasement (>180°) of a short segment of the hepatic artery

OR

Anatomic variation of the visceral arteries with vascularization of the liver or mesentery via collaterals which need to be ligated during tumor resection (e.g. gastroduodenal artery), as shown on CT or MRI

OR

High-grade stenosis or occlusion of either the celiac trunk or the superior mesenteric artery with vascularization of the liver or mesentery via collaterals which need to be ligated during tumor resection (e.g. gastroduodenal artery), as shown on CT or MRI, which is not amenable to endovascular revascularization

* Invasion of the portal or superior mesenteric vein may be present, but must be considered resectable (involvement with distortion or narrowing of the vein or occlusion of the vein with suitable vessel proximal and distal, allowing for safe resection and replacement) according to National Comprehensive Cancer Network (NCCN) and International Study Group of Pancreatic Surgery (ISGPS) criteria (11, 12)
* Provision of written informed consent prior to performance of study-specific procedures or assessments and willingness to comply with treatment and follow-up

Exclusion Criteria

* Histologically proven peritoneal carcinomatosis (biopsies of macroscopically suspicious findings must be taken at the beginning of the operation and be analyzed immediately by fresh frozen section)
* Histologically proven distant metastatic disease
* Co-morbidities, organ function or physical status precluding visceral debranching or intensive neoadjuvant combination chemotherapy, as judged by the treating physicians
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with the patient's safety, provision of informed consent, or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of visceral debranching | Six weeks
  Proportion of patients proceeding to neoadjuvant chemotherapy (at least one dose administered within six weeks from the debranching procedure) among all patients undergoing visceral debranching

SECONDARY OUTCOMES:
Completion of therapy | Three months
  Proportion of patients proceeding to attempted tumor resection among all patients undergoing visceral debranching
Completeness of resection | Three months
  Proportion of patients with clear resection margins (R0) upon pancreatic cancer resection following visceral debranching and neoadjuvant chemotherapy among all patients undergoing visceral debranching
Perioperative morbidity (visceral debranching) | Four weeks
  Perioperative in-hospital morbidity associated with the visceral debranching procedure, measured according to the Clavien-Dindo-Classification of surgical complications
Perioperative morbidity (pancreatic cancer resection) | Four weeks
  Perioperative in-hospital morbidity associated with pancreatic cancer resection, measured according to the Clavien-Dindo-Classification of surgical complications
Toxicity of chemotherapy | Three months
  Toxicity during neoadjuvant chemotherapy, measured according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Progression-free survival | Three years
  Time between time between first diagnosis, which is assumed to be equivalent to study enrolment, and documented progression. For patients who are not resected, progression-free survival will be defined as zero
Recurrence-free survival | Three years
  Time between resection and the appearance of local recurrence, peritoneal carcinomatosis, or distant metastases. For patients who are not resected, recurrence-free survival will be defined as zero
Overall survival | Three years
  Time between time between first diagnosis, which is assumed to be equivalent to study enrolment, and death, independent of the cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Kleeff, MD, Principal Investigator — Martin-Luther-Universität Halle-Wittenberg
Locations (3):
- Germany (3):
  - University Hospital, Dpt. of Visceral, Vascular and Endocrine Surgery, Halle
  - University Hospital, Heidelberg
  - University Hospital, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ronellenfitsch U, Michalski CW, Michl P, Krug S, Ukkat J, Kleeff J. Pre-operative/Neoadjuvant Therapy and Vascular Debranching Followed by Resection for Locally Advanced Pancreatic Cancer (PREVADER): Clinical Feasibility Trial. Front Med (Lausanne). 2021 May 24;8:588375. doi: 10.3389/fmed.2021.588375. eCollection 2021. PMID 34109185